CLINICAL TRIAL: NCT00097591
Title: A Comparison of CS-747 and Clopidogrel in Acute Coronary Syndrome Subjects Who Are to Undergo Percutaneous Coronary Intervention
Brief Title: A Comparison of Prasugrel (CS-747) and Clopidogrel in Acute Coronary Syndrome Subjects Who Are to Undergo Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Chief Medical Officer, Eli LIlly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8695; H7T-MC-TAAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Arteriosclerosis; Acute Coronary Syndromes
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): Oral loading dose of six 10 mg prasugrel tablets and four placebo tablets matched to clopidogrel, followed by an oral maintenance dose of prasugrel one 10 mg tablet and one placebo tablet matched to clopidogrel once daily
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Oral loading dose of four 75 mg clopidogrel tablets and six placebo tablets matched to prasugrel, followed by an oral maintenance dose of one 75 mg clopidogrel tablet and one placebo tablet matched to prasugrel once daily
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Administered orally
  Other Names: CS-747; LY640315; Effient; Efient
  Arms: Prasugrel
Drug: Clopidogrel — Administered orally
  Arms: Clopidogrel

SUMMARY:
The sponsors of this investigational drug are developing prasugrel (also known as CS-747) as a possible treatment for patients with acute coronary syndrome (heart attack or chest pain) who need, or are expected to need, a percutaneous coronary intervention (PCI; also called a balloon angioplasty). Prasugrel was compared with Clopidogrel to determine which drug is better at reducing deaths, future heart attacks, or stroke.

ELIGIBILITY:
Inclusion Criteria:

* A person who has been diagnosed with acute coronary syndrome and is to undergo a percutaneous coronary intervention.
* A person who is of the legal age of 18 and is mentally competent to provide a signed written informed consent.
* If a woman is of childbearing potential (i.e., before menopause), she must test negative for pregnancy and agree to use a reliable method of birth control.

Exclusion Criteria:

* A person who has had an ischemic stroke within the last 3 months or a hemorrhagic stroke at any time in the past.
* A person who has active internal bleeding or has a history of a bleeding disorder.
* Individuals who are at an increased risk of bleeding based on laboratory criteria evaluated by the treatment physician or on medication that can cause bleeding.
* A person who has liver disease; for example, cirrhosis.
* A person who has a condition such as alcoholism, mental illness, or is drug dependent.
* A person who has cardiogenic shock, a refractory ventricular arrhythmia, or congestive heart failure (class IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13619 (Actual)
Dates: Start 2004-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For more information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Global Quintiles Study Line (1-866-615-4672) or speak with your physician, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Pride YB, Tung P, Mohanavelu S, Zorkun C, Wiviott SD, Antman EM, Giugliano R, Braunwald E, Gibson CM; TIMI Study Group. Angiographic and clinical outcomes among patients with acute coronary syndromes presenting with isolated anterior ST-segment depression: a TRITON-TIMI 38 (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition With Prasugrel-Thrombolysis In Myocardial Infarction 38) substudy. JACC Cardiovasc Interv. 2010 Aug;3(8):806-11. doi: 10.1016/j.jcin.2010.05.012. PMID 20723851
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Scirica BM, Bergmark BA, Morrow DA, Antman EM, Bonaca MP, Murphy SA, Sabatine MS, Braunwald E, Wiviott SD. Nonculprit Lesion Myocardial Infarction Following Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome. J Am Coll Cardiol. 2020 Mar 17;75(10):1095-1106. doi: 10.1016/j.jacc.2019.12.067. PMID 32164882
- [Derived] Cowper PA, Knight JD, Davidson-Ray L, Peterson ED, Wang TY, Mark DB; TRANSLATE-ACS Investigators. Acute and 1-Year Hospitalization Costs for Acute Myocardial Infarction Treated With Percutaneous Coronary Intervention: Results From the TRANSLATE-ACS Registry. J Am Heart Assoc. 2019 Apr 16;8(8):e011322. doi: 10.1161/JAHA.118.011322. PMID 30975005
- [Derived] Udell JA, Braunwald E, Antman EM, Murphy SA, Montalescot G, Wiviott SD. Prasugrel versus clopidogrel in patients with ST-segment elevation myocardial infarction according to timing of percutaneous coronary intervention: a TRITON-TIMI 38 subgroup analysis (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition with Prasugrel-Thrombolysis In Myocardial Infarction 38). JACC Cardiovasc Interv. 2014 Jun;7(6):604-12. doi: 10.1016/j.jcin.2014.01.160. PMID 24947719
- [Derived] Kohli P, Udell JA, Murphy SA, Cannon CP, Antman EM, Braunwald E, Wiviott SD. Discharge aspirin dose and clinical outcomes in patients with acute coronary syndromes treated with prasugrel versus clopidogrel: an analysis from the TRITON-TIMI 38 study (trial to assess improvement in therapeutic outcomes by optimizing platelet inhibition with prasugrel-thrombolysis in myocardial infarction 38). J Am Coll Cardiol. 2014 Jan 28;63(3):225-32. doi: 10.1016/j.jacc.2013.09.023. Epub 2013 Oct 16. PMID 24140678
- [Derived] Goodnough LT, Smith PK, Levy JH, Poston RS, Short MA, Weerakkody GJ, LeNarz LA. Transfusion outcomes in patients undergoing coronary artery bypass grafting treated with prasugrel or clopidogrel: TRITON-TIMI 38 retrospective data analysis. J Thorac Cardiovasc Surg. 2013 Apr;145(4):1077-1082.e4. doi: 10.1016/j.jtcvs.2012.07.059. Epub 2012 Sep 17. PMID 22995726
- [Derived] Smith PK, Goodnough LT, Levy JH, Poston RS, Short MA, Weerakkody GJ, Lenarz LA. Mortality benefit with prasugrel in the TRITON-TIMI 38 coronary artery bypass grafting cohort: risk-adjusted retrospective data analysis. J Am Coll Cardiol. 2012 Jul 31;60(5):388-96. doi: 10.1016/j.jacc.2012.03.030. Epub 2012 May 23. PMID 22633653
- [Derived] Bonaca MP, Wiviott SD, Braunwald E, Murphy SA, Ruff CT, Antman EM, Morrow DA. American College of Cardiology/American Heart Association/European Society of Cardiology/World Heart Federation universal definition of myocardial infarction classification system and the risk of cardiovascular death: observations from the TRITON-TIMI 38 trial (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition With Prasugrel-Thrombolysis in Myocardial Infarction 38). Circulation. 2012 Jan 31;125(4):577-83. doi: 10.1161/CIRCULATIONAHA.111.041160. Epub 2011 Dec 23. PMID 22199016
- [Derived] Hochholzer W, Wiviott SD, Antman EM, Contant CF, Guo J, Giugliano RP, Dalby AJ, Montalescot G, Braunwald E. Predictors of bleeding and time dependence of association of bleeding with mortality: insights from the Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition With Prasugrel--Thrombolysis in Myocardial Infarction 38 (TRITON-TIMI 38). Circulation. 2011 Jun 14;123(23):2681-9. doi: 10.1161/CIRCULATIONAHA.110.002683. Epub 2011 May 23. PMID 21606391
- [Derived] Mahoney EM, Wang K, Arnold SV, Proskorovsky I, Wiviott S, Antman E, Braunwald E, Cohen DJ. Cost-effectiveness of prasugrel versus clopidogrel in patients with acute coronary syndromes and planned percutaneous coronary intervention: results from the trial to assess improvement in therapeutic outcomes by optimizing platelet inhibition with Prasugrel-Thrombolysis in Myocardial Infarction TRITON-TIMI 38. Circulation. 2010 Jan 5;121(1):71-9. doi: 10.1161/CIRCULATIONAHA.109.900704. Epub 2009 Dec 21. PMID 20026770
- [Derived] Pride YB, Wiviott SD, Buros JL, Zorkun C, Tariq MU, Antman EM, Braunwald E, Gibson CM; TIMI Study Group. Effect of prasugrel versus clopidogrel on outcomes among patients with acute coronary syndrome undergoing percutaneous coronary intervention without stent implantation: a TRial to assess Improvement in Therapeutic Outcomes by optimizing platelet inhibitioN with prasugrel (TRITON)-Thrombolysis in Myocardial Infarction (TIMI) 38 substudy. Am Heart J. 2009 Sep;158(3):e21-6. doi: 10.1016/j.ahj.2009.06.021. PMID 19699846
- [Derived] Montalescot G, Wiviott SD, Braunwald E, Murphy SA, Gibson CM, McCabe CH, Antman EM; TRITON-TIMI 38 investigators. Prasugrel compared with clopidogrel in patients undergoing percutaneous coronary intervention for ST-elevation myocardial infarction (TRITON-TIMI 38): double-blind, randomised controlled trial. Lancet. 2009 Feb 28;373(9665):723-31. doi: 10.1016/S0140-6736(09)60441-4. PMID 19249633
- [Derived] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Derived] Wiviott SD, Braunwald E, Angiolillo DJ, Meisel S, Dalby AJ, Verheugt FW, Goodman SG, Corbalan R, Purdy DA, Murphy SA, McCabe CH, Antman EM; TRITON-TIMI 38 Investigators. Greater clinical benefit of more intensive oral antiplatelet therapy with prasugrel in patients with diabetes mellitus in the trial to assess improvement in therapeutic outcomes by optimizing platelet inhibition with prasugrel-Thrombolysis in Myocardial Infarction 38. Circulation. 2008 Oct 14;118(16):1626-36. doi: 10.1161/CIRCULATIONAHA.108.791061. Epub 2008 Aug 31. PMID 18757948
- [Derived] Antman EM, Wiviott SD, Murphy SA, Voitk J, Hasin Y, Widimsky P, Chandna H, Macias W, McCabe CH, Braunwald E. Early and late benefits of prasugrel in patients with acute coronary syndromes undergoing percutaneous coronary intervention: a TRITON-TIMI 38 (TRial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet InhibitioN with Prasugrel-Thrombolysis In Myocardial Infarction) analysis. J Am Coll Cardiol. 2008 May 27;51(21):2028-33. doi: 10.1016/j.jacc.2008.04.002. PMID 18498956
- [Derived] Wiviott SD, Braunwald E, McCabe CH, Horvath I, Keltai M, Herrman JP, Van de Werf F, Downey WE, Scirica BM, Murphy SA, Antman EM; TRITON-TIMI 38 Investigators. Intensive oral antiplatelet therapy for reduction of ischaemic events including stent thrombosis in patients with acute coronary syndromes treated with percutaneous coronary intervention and stenting in the TRITON-TIMI 38 trial: a subanalysis of a randomised trial. Lancet. 2008 Apr 19;371(9621):1353-63. doi: 10.1016/S0140-6736(08)60422-5. Epub 2008 Apr 2. PMID 18377975
- [Derived] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Acute Coronary Syndromes (ACS) includes subjects presenting with unstable angina (UA), non-ST-segment elevation myocardial infarction (NSTEMI), and ST-segment elevation myocardial infarction (STEMI).
Period: Overall Study
Arm/Group | Prasugrel | Clopidogrel
Started | 6813 (7 subjects randomized but not analyzed due to an incomplete informed consent document) | 6795 (4 subjects randomized but not analyzed due to an incomplete informed consent document)
Completed | 6403 | 6401
Not Completed | 410 | 394
Not completed — Withdrawal of consent | 342 | 323
Not completed — Less than 6 months on study drug | 9 | 7
Not completed — Unable to attend termination visit | 53 | 51
Not completed — Lost to follow up | 6 | 10
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Total
Number analyzed (Participants) | 6813 | 6795 | 13608
Age Continuous [Mean (Standard Deviation); unit: years] | 60.9 (11.2) | 60.9 (11.4) | 60.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1705 | 1818 | 3523
  Male | 5108 | 4977 | 10085
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 6263 | 6274 | 12537
  African | 205 | 187 | 392
  Hispanic | 269 | 256 | 525
  Asian | 60 | 64 | 124
  Other | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  North America | 2164 | 2146 | 4310
  South America | 270 | 264 | 534
  Europe | 3436 | 3439 | 6875
  Middle East | 606 | 613 | 1219
  Africa | 204 | 200 | 404
  Pacifica | 133 | 133 | 266

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reaching the Composite Endpoint of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), or Nonfatal Stroke
Description: The endpoint in this measure is a combination of CV death, nonfatal MI, or nonfatal stroke. The data is presented by the study population, which is represented as follows: 1) subjects who presented with unstable angina and non-ST-segment elevation myocardial infarction (UA/NSTEMI), 2) subjects who presented with ST segment elevation myocardial infarction (STEMI), and 3) all subjects with acute coronary syndromes (ACS) (i.e. all subjects with UA/NSTEMI or STEMI).
Time Frame: Randomization up to 15 months
Population: Intention-to-treat (ITT) population consisting of all subjects with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) who may or may not have received study drug
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6813 | 6795
Participants
  UA/NSTEMI (n=5044, n=5030) | 469 | 565
  STEMI (n=1769, n=1765) | 174 | 216
  All ACS (n=6813, n=6795) | 643 | 781
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; For UA/NSTEMI population; Test type: Superiority or Other; p = 0.002, Gehan-Wilcoxon — The primary outcome measure was analyzed first in the UA/NSTEMI population, followed by All ACS subjects, followed by the STEMI population; Hazard Ratio (HR) = 0.820, 95% CI 2-sided [0.726 to 0.927]
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; For STEMI population; Test type: Superiority or Other; p = 0.019, Gehan-Wilcoxon; Hazard Ratio (HR) = 0.793, 95% CI 2-sided [0.649 to 0.968]
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; For All ACS population; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.812, 95% CI 2-sided [0.732 to 0.902]

2. Secondary Outcome: Number of Treated Subjects With Non-Coronary Artery Bypass Graft (CABG) Related Thrombolysis In Myocardial Infarction (TIMI) Study Group Major and Minor Bleeding Events
Description: TIMI classification for major and minor bleeding in the subset of subjects who did not undergo a coronary artery bypass operation (CABG) were defined as follows: Major bleeding: any intracranial hemorrhage (ICH) OR any clinically overt bleeding (including bleeding evident on imaging studies) associated with a fall in hemoglobin (Hgb) of ≥5 grams/deciliter (gm/dL)from baseline. Minor Bleeding: any clinically overt bleeding associated with a fall in Hgb of ≥3 gm/dL but <5 gm/dL from baseline. Major bleeding events were further examined as events that were deemed life threatening and/or fatal.
Time Frame: First dose of study drug up to 15 months (while at risk)
Population: Treated subjects with adverse events were considered "at risk" from the first dose of study drug up through 7 days after permanent study drug discontinuation, or the subjects' discontinuation visit; or from randomization through 464 days, whichever is earlier. Adverse events classified as "study drug related" were included in the "at risk" set.
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6741 | 6716
Participants
  TIMI Major or Minor Bleeding | 303 | 231
  TIMI Major Bleeding | 146 | 111
  TIMI Major Bleeding - Life-threatening (LT) | 85 | 56
  LT - Fatal | 21 | 5
  LT - Symptomatic intracranial hemorrage (ICH) | 19 | 17
  LT - Requiring inotropes | 21 | 8
  LT - Requiring surgical intervention | 19 | 19
  LT - Requiring transfusion (>=4 units) | 45 | 30
  TIMI Minor Bleeding | 164 | 125
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; For non-CABG TIMI Major or Minor Bleeding; Test type: Superiority or Other; p = 0.002, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.314, 95% CI 2-sided [1.107 to 1.559]
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; For non-CABG TIMI Major Bleeding; Test type: Superiority or Other; p = 0.029, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.315, 95% CI 2-sided [1.028 to 1.683]
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - Life-threatening events (LT); Test type: Superiority or Other; p = 0.015, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.517, 95% CI 2-sided [1.083 to 2.126]
Statistical Analysis 4: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - LT - Fatal; Test type: Superiority or Other; p = 0.002, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 4.191, 95% CI 2-sided [1.1580 to 11.113]
Statistical Analysis 5: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - LT - Symptomatic intracranial hemorrage (ICH); Test type: Superiority or Other; p = 0.736, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.119, 95% CI 2-sided [0.582 to 2.152]
Statistical Analysis 6: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - LT - Requiring inotropes; Test type: Superiority or Other; p = 0.016, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 2.617, 95% CI 2-sided [1.159 to 5.908]
Statistical Analysis 7: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - LT - Requiring surgical intervention; Test type: Superiority or Other; p = 0.995, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.998, 95% CI 2-sided [0.528 to 1.885]
Statistical Analysis 8: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Major Bleeding - LT - Requiring transfusion (>=4 units); Test type: Superiority or Other; p = 0.084, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.499, 95% CI 2-sided [0.945 to 2.379]
Statistical Analysis 9: Comparison: Prasugrel vs Clopidogrel; For the subset of non-CABG TIMI Minor Bleeding; Test type: Superiority or Other; p = 0.022, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 1.313, 95% CI 2-sided [1.040 to 1.656]

3. Secondary Outcome: Number of Subjects Reaching the Composite Endpoint of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), or Urgent Target Vessel Revascularization (UTVR)
Description: The endpoint in this measure is a combination of CV death, nonfatal MI, or UTVR. Results are reported for the All ACS subject population for the 30 and 90 day periods.
Time Frame: Randomization to 30 days; randomization to 90 days
Population: Intention-to-treat (ITT) population consisting of all randomized All ACS subjects who may or may not have received study drug.
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6813 | 6795
Participants
  All ACS (Through 30 days) | 399 | 504
  All ACS (Through 90 days) | 472 | 588
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Through 30 days; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.784, 95% CI 2-sided [0.688 to 0.894]
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; Through 90 days; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.703 to 0.896]

4. Secondary Outcome: Number of Subjects Reaching the Composite Endpoint of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), or Nonfatal Stroke
Description: The endpoint in this measure is a combination of CV death, nonfatal MI, or nonfatal stroke. Results are reported for the All ACS population for the 30 and 90 day periods.
Time Frame: Randomization to 30 days; randomization to 90 days
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6813 | 6795
Participants
  All ACS (Through 30 days) | 389 | 502
  All ACS (Through 90 days) | 462 | 573
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Through 30 days; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.767, 95% CI 2-sided [0.672 to 0.876]
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; Through 90 days; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.705 to 0.901]

5. Secondary Outcome: Number of Subjects Reaching the Composite Endpoint of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, or Rehospitalization for Cardiac Ischemic Events
Description: The endpoint in this measure is a combination of CV death, nonfatal MI, nonfatal stroke, or rehospitalization for cardiac ischemic events. Results are reported for the All ACS population.
Time Frame: Randomization up to 15 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6813 | 6795
Participants | 797 | 938
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.838, 95% CI 2-sided [0.762 to 0.921]

6. Secondary Outcome: Number of Subjects Reaching the Composite Endpoint of All-Cause Death, Nonfatal Myocardial Infarction (MI), or Nonfatal Stroke
Description: The endpoint in this measure is a combination of all-cause death, nonfatal MI, or nonfatal stroke. Results are reported for the All ACS population.
Time Frame: Randomization up to 15 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 6813 | 6795
Participants | 692 | 822
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Log Rank; Clinical presentation, UA/NSTEMI versus STEMI, was used as a stratification factor; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.751 to 0.919]

ADVERSE EVENTS:
Arm/Group | Prasugrel | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 1731/6741 | 1675/6716
Other Adverse Events (participants affected / at risk) | 5217/6741 | 5187/6716
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=6741) | Clopidogrel (N=6716)
Anaemia (Blood and lymphatic system disorders) | 39 (39) | 34 (35)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 15 (15)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 1 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 85 (87) | 86 (95)
Angina unstable (Cardiac disorders) | 25 (27) | 37 (39)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 3 (4)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 50 (51) | 52 (56)
Atrial flutter (Cardiac disorders) | 12 (12) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 5 (5)
Atrioventricular block third degree (Cardiac disorders) | 11 (11) | 11 (11)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 14 (14) | 11 (11)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 10 (10) | 10 (12)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 22 (24) | 41 (42)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 3 (4)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 46 (48) | 47 (48)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pseudoaneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 5 (5) | 4 (4)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 13 (14) | 8 (8)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 4 (4) | 2 (2)
Coronary artery aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 14 (14) | 17 (17)
Coronary artery dissection (Cardiac disorders) | 5 (5) | 11 (11)
Coronary artery occlusion (Cardiac disorders) | 8 (8) | 7 (7)
Coronary artery perforation (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery restenosis (Cardiac disorders) | 107 (118) | 111 (118)
Coronary artery stenosis (Cardiac disorders) | 52 (54) | 64 (65)
Coronary artery thrombosis (Cardiac disorders) | 2 (2) | 2 (4)
Dressler's syndrome (Cardiac disorders) | 4 (4) | 2 (2)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 1 (1)
In-stent arterial restenosis (Cardiac disorders) | 0 (0) | 1 (1)
Interventricular septum rupture (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 9 (9) | 4 (4)
Ischaemic cardiomyopathy (Cardiac disorders) | 6 (6) | 3 (3)
Left ventricular failure (Cardiac disorders) | 1 (2) | 4 (4)
Low cardiac output syndrome (Cardiac disorders) | 3 (3) | 2 (2)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 6 (6) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 12 (13) | 17 (17)
Myocardial rupture (Cardiac disorders) | 0 (0) | 2 (2)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Papillary muscle disorder (Cardiac disorders) | 0 (0) | 1 (1)
Papillary muscle rupture (Cardiac disorders) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 8 (11) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 5 (5) | 7 (8)
Pericarditis (Cardiac disorders) | 3 (4) | 8 (9)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (2)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 5 (5)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 2 (2) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 8 (10) | 5 (6)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Torsade de pointes (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 6 (6) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 18 (19) | 25 (25)
Ventricular flutter (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular septal defect acquired (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 24 (27) | 25 (30)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Laryngocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Auricular perichondritis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Vestibular neuronitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Cataract (Eye disorders) | 4 (4) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 4 (4) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 1 (1)
Hyphaema (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (2) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (3) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal haematoma (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 10 (10)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 7 (7)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 8 (8)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 8 (8) | 6 (6)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5 (5) | 5 (5)
Gastritis (Gastrointestinal disorders) | 7 (7) | 7 (8)
Gastritis erosive (Gastrointestinal disorders) | 7 (7) | 3 (3)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 91 (95) | 55 (61)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 11 (11)
Gastrooesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 6 (6) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Intestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (8) | 10 (11)
Mallory-weiss syndrome (Gastrointestinal disorders) | 3 (3) | 2 (2)
Melaena (Gastrointestinal disorders) | 6 (6) | 6 (6)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 6 (6) | 3 (4)
Pancreatitis acute (Gastrointestinal disorders) | 5 (5) | 5 (5)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Polyp colorectal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 11 (11) | 5 (5)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Retroperitoneal haematoma (Gastrointestinal disorders) | 5 (5) | 4 (4)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 15 (16) | 9 (9)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 15 (16) | 8 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abasia (General disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 4 (4) | 3 (3)
Catheter site haemorrhage (General disorders) | 1 (2) | 1 (1)
Chest discomfort (General disorders) | 7 (7) | 7 (8)
Chest pain (General disorders) | 91 (98) | 73 (78)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (General disorders) | 1 (1) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 3 (3)
Ischaemic ulcer (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-organ disorder (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 138 (155) | 167 (179)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Puncture site haemorrhage (General disorders) | 30 (30) | 18 (18)
Pyrexia (General disorders) | 12 (13) | 6 (6)
Submandibular mass (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 2 (2)
Vessel puncture site haematoma (General disorders) | 21 (21) | 14 (14)
Vessel puncture site haemorrhage (General disorders) | 13 (13) | 10 (10)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 7 (7)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 10 (10) | 13 (13)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 2 (2)
Anaphylactic shock (Immune system disorders) | 2 (2) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Hypersensitivity (Immune system disorders) | 3 (3) | 2 (3)
Polyarteritis nodosa (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 5 (5) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5)
Bronchitis acute (Infections and infestations) | 9 (9) | 3 (3)
Bronchitis chronic (Infections and infestations) | 0 (0) | 3 (3)
Bronchopneumonia (Infections and infestations) | 5 (5) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 11 (12) | 6 (6)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 8 (10) | 5 (5)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (10) | 6 (6)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Localised infection (Infections and infestations) | 0 (0) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 2 (2)
Mediastinitis (Infections and infestations) | 0 (0) | 3 (3)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Perianal abscess (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 43 (45) | 52 (54)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 1 (1)
Pyothorax (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 8 (8) | 9 (9)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 4 (4) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6)
Urinary tract infection (Infections and infestations) | 15 (17) | 19 (19)
Urosepsis (Infections and infestations) | 6 (6) | 3 (3)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 4 (4) | 3 (3)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 3 (3)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 0 (0)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Eyeball rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure of implant (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (12) | 12 (12)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hepatic trauma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 17 (18) | 7 (7)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 20 (20) | 8 (8)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Angiogram (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Cardiac enzymes increased (Investigations) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 2 (2) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1)
Electrocardiogram st segment elevation (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 10 (10) | 6 (6)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Prostate examination abnormal (Investigations) | 2 (2) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 3 (3)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 14 (14) | 9 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 15 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell carcinoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral t-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (2)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 1 (2)
Carotid artery stenosis (Nervous system disorders) | 18 (19) | 10 (12)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 5 (5) | 2 (2)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 3 (3)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 8 (8)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 0 (0) | 1 (1)
Global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 5 (5) | 4 (4)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 4 (4)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Iiird nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 2 (3)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Periodic limb movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 11 (11) | 8 (8)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 35 (35) | 29 (31)
Syncope vasovagal (Nervous system disorders) | 4 (4) | 4 (4)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 16 (17) | 22 (23)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 7 (7)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 5 (5) | 5 (5)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 3 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 3 (3) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Crush syndrome (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 27 (31) | 12 (14)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 7 (7) | 2 (2)
Nephropathy (Renal and urinary disorders) | 1 (1) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 15 (15) | 17 (17)
Renal failure acute (Renal and urinary disorders) | 22 (22) | 12 (12)
Renal failure chronic (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal impairment (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 5 (5)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (8)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 13 (13)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 21 (21)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 22 (23)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 31 (38) | 27 (29)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 6 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Dental operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Eye operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 2 (2)
Open reduction of fracture (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 1 (1)
Thrombectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 2 (2)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 4 (4) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Arterial restenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 2 (2) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 3 (3)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 13 (13) | 10 (10)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 2 (3) | 4 (5)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 4 (4) | 3 (3)
Haematoma (Vascular disorders) | 16 (16) | 17 (17)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 8 (8) | 5 (5)
Hypertension (Vascular disorders) | 17 (17) | 16 (16)
Hypertensive crisis (Vascular disorders) | 13 (13) | 15 (15)
Hypertensive emergency (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 15 (15) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 3 (3) | 5 (5)
Iliac artery stenosis (Vascular disorders) | 2 (2) | 6 (7)
Intermittent claudication (Vascular disorders) | 5 (5) | 3 (4)
Ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (5) | 3 (3)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 3 (4)
Peripheral vascular disorder (Vascular disorders) | 8 (8) | 11 (11)
Reperfusion injury (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 25 (26) | 26 (26)
Vascular stenosis (Vascular disorders) | 0 (0) | 1 (1)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Wound haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=6741) | Clopidogrel (N=6716)
Angina pectoris (Cardiac disorders) | 302 (340) | 334 (382)
Nausea (Gastrointestinal disorders) | 308 (327) | 290 (306)
Chest pain (General disorders) | 690 (818) | 643 (771)
Fatigue (General disorders) | 249 (261) | 324 (339)
Contusion (Injury, poisoning and procedural complications) | 464 (529) | 262 (302)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 325 (325) | 325 (325)
Back pain (Musculoskeletal and connective tissue disorders) | 336 (358) | 304 (326)
Dizziness (Nervous system disorders) | 271 (298) | 300 (325)
Headache (Nervous system disorders) | 372 (402) | 353 (388)
Cough (Respiratory, thoracic and mediastinal disorders) | 264 (277) | 274 (281)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 319 (339) | 284 (295)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 398 (480) | 204 (251)
Coronary revascularisation (Surgical and medical procedures) | 313 (346) | 389 (427)
Percutaneous coronary intervention (Surgical and medical procedures) | 668 (748) | 690 (779)
Haematoma (Vascular disorders) | 426 (474) | 357 (378)
Hypertension (Vascular disorders) | 490 (495) | 460 (468)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days